CLINICAL TRIAL: NCT03911544
Title: Does Bispectral Index Improve Surgical Conditions During Fast Track Gynecological Benign Laparoscopies
Brief Title: Bispectral Index and Surgical Field
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Elena Crescioli, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20190006
Record Dates: First submitted 2019-04-06; First posted 2019-04-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Consciousness Monitors; Laparoscopy
Keywords: Neuromuscular Agents; Bispectral Index

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA anesthesia with BIS monitoring (Active Comparator): The depth of anesthesia will be adjusted with the help of BIS monitoring.
  Interventions: Device: BIS monitor
- TIVA anesthesia without BIS monitoring (No Intervention): The depth of anesthesia will adjusted as in standard practice (clinical signs of poor anesthesia such as increase in blood pressure and/or heart rate, tearing and profuse sweating)

INTERVENTIONS:
Device: BIS monitor — Participants allocated to the intervention group will receive TIVA anesthesia adjusted by the BIS monitoring in addition to clinical signs of poor anesthesia.
  Arms: TIVA anesthesia with BIS monitoring

SUMMARY:
This study investigates whether BIS monitor assisted anesthesia improves surgical space conditions during gynecological benign laparoscopic procedures.

Half of participants will receive BIS monitor assisted anesthesia, while the other half will receive anesthesia without BIS monitor.

DETAILED DESCRIPTION:
General Anesthesia includes hypnosis/unconsciousness, amnesia, analgesia, muscle relaxation and autonomic and sensory blockade of responses to noxious stimulation.

Depth of anesthesia in standard practice is controlled by monitoring equipment such as blood pressure (BP), heart rate (HR), train of four ratio (TOF) and by clinical signs such as profuse sweating, tearing, cough and movements.

BIS can be used as additional tool to monitor and manage anesthesia. BIS is an empirically derived scale for measuring brain electrical activity. It computes an index between 0 and 100, whereas 0 corresponds to "no detectable brain electrical activity" (flatline EEG) and 100 to awake state. A patient is considered to be appropriately anesthetized when the BIS' value is between 40 and 60.

ELIGIBILITY:
Inclusion Criteria:

* Women aged > 18 years
* American Society of Anesthesiology (ASA) physical status 1 or 2
* Legally competent

Exclusion Criteria:

* Age < 18 years
* ASA physical status ≥3
* Renal and/or lever disease
* Relevant allergies towards anesthetics
* Cancer surgery
* No informed consent or inability to give that

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Proportion of optimal surgical field score | up to 12 hours
  score 1 on a scale 1-4 (higher values represent a better outcome)

SECONDARY OUTCOMES:
Administration of neuromuscular block | up to 12 hours
  Total amount of neuromuscolar block given during anesthesia, expressed in milligrams
Amount of anesthetics, narcotic analgesics and other adjuvants | up to 12 hours
  Registration is in milligrams
BIS values (continues) | up to 12 hours
  continues values
Event of PONV (postoperative nausea and vomiting) and antiemetic administration in post-anesthesia care unit (PACU) | 1 day
  Registration of the drugs in in milligrams
Amount of analgesics administered in PACU | 1 day
  Registration is in milligrams

CONTACTS AND LOCATIONS:
Overall Officials: Elena Crescioli, M.D., Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Result] Song D, Joshi GP, White PF. Titration of volatile anesthetics using bispectral index facilitates recovery after ambulatory anesthesia. Anesthesiology. 1997 Oct;87(4):842-8. doi: 10.1097/00000542-199710000-00018. PMID 9357886
- [Result] Ahmad S, Yilmaz M, Marcus RJ, Glisson S, Kinsella A. Impact of bispectral index monitoring on fast tracking of gynecologic patients undergoing laparoscopic surgery. Anesthesiology. 2003 Apr;98(4):849-52. doi: 10.1097/00000542-200304000-00010. PMID 12657845
- [Result] Kamal NM, Omar SH, Radwan KG,Youssef A. Bispectral Index Monitoring Tailors Clinical Anesthetic Delivery and Reduces Anesthetic Drug Consumption. Journal of Medical Sciences, 9: 10-16, 2009
- [Result] Madsen MV, Staehr-Rye AK, Claudius C, Gatke MR. Is deep neuromuscular blockade beneficial in laparoscopic surgery? Yes, probably. Acta Anaesthesiol Scand. 2016 Jul;60(6):710-6. doi: 10.1111/aas.12698. Epub 2016 Feb 10. PMID 26864853
- [Result] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Result] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Result] Madsen MV, Gatke MR, Springborg HH, Rosenberg J, Lund J, Istre O. Optimising abdominal space with deep neuromuscular blockade in gynaecologic laparoscopy--a randomised, blinded crossover study. Acta Anaesthesiol Scand. 2015 Apr;59(4):441-7. doi: 10.1111/aas.12493. Epub 2015 Mar 1. PMID 25789421
- [Derived] Crescioli E, Thyrrestrup PS, Almas T. Bispectral Index and Surgical Space Conditions in Day Surgery Benign Gynecological Laparoscopies: A Double-Blinded Randomized Clinical Trial. Anesthesiol Res Pract. 2025 Feb 23;2025:4558323. doi: 10.1155/anrp/4558323. eCollection 2025. PMID 40026610
- See also: D. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. — https://www.bmj.com/content/340/bmj.c332